CLINICAL TRIAL: NCT00286754
Title: A Behavioral Intervention to Improve Hypertension Control in Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 04-170
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension
Keywords: Hypertension; Behavior modification; Randomized controlled trial; Treatment effectiveness; Telemedicine; Prevention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stage-matched intervention (SMI) (Experimental): Stage-matched intervention (SMI)
  Interventions: Behavioral: SMI; Behavioral: HEI; Behavioral: UC
- Health Education Intervention (HEI) (Active Comparator): Health Education Intervention (HEI)
  Interventions: Behavioral: SMI; Behavioral: HEI; Behavioral: UC
- Usual Care (UC) (No Intervention): Usual Care (UC)

INTERVENTIONS:
Behavioral: SMI — Stage-matched intervention
  Arms: Stage-matched intervention (SMI)
Behavioral: HEI — Health Education Intervention
  Arms: Stage-matched intervention (SMI)
Behavioral: UC — Usual Care
  Arms: Stage-matched intervention (SMI)
Behavioral: SMI — Stage-matched intervention
  Arms: Health Education Intervention (HEI)
Behavioral: HEI — Health Education Intervention
  Arms: Health Education Intervention (HEI)
Behavioral: UC — Usual Care
  Arms: Health Education Intervention (HEI)

SUMMARY:
The purpose of this study is to determine whether a stage-matched intervention (SMI) will lower BP and improve treatment adherence compared to usual care (UC) or a health education intervention (HEI) in veterans with uncontrolled BP. The study will also examine the effect of SMI on patient's health-related quality of life, satisfaction, acceptability and determine its cost-effectiveness.

DETAILED DESCRIPTION:
We propose a randomized controlled trial to evaluate the effect of telephone-delivered interventions (SMI and HEI) to improve BP control.

Veterans with uncontrolled hypertension (n=533) will be randomized equally to 3 groups: 1) The SMI will use the Transtheoretical model (TTM) as the unifying framework. Veterans will receive TTM stage-matched counseling for exercise, diet, and medications via monthly counseling sessions. A social worker (SW) will assess each participant's behavior and deliver the appropriate tailored SMI based on their stage of change, decisional balance, self-efficacy and the skills model questions. 2) The HEI group receives monthly telephone calls by a SW during which they will receive education about hypertension management. 3) The UC group participates in all the in-person visits but does not receive monthly calls.

There will be an initial 6-month active intervention phase followed by a 6 month monitoring phase to assess sustainability. All participants will visit the VAMC's at baseline and at 3, 6, and 12 months. Outcomes of interest include BP; adherence (to diet, exercise and medications); quality of life; satisfaction; acceptability; cost and cost-effectiveness. Patients will be blinded to which of the intervention arms (SMI or HEI) they are in, SW's will be blinded to patient's BP and staff measuring outcomes will be blinded to study assignment. The study will be analyzed using longitudinal data analysis methods using an intention to treat strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving continuity of care in the outpatient clinics will be eligible. This will be operationalized as 2 visits in the previous year.
* Adults (= 21 years) with hypertension, on antihypertensive medication for = 1 year, and who have current uncontrolled BP will be enrolled.

Patients with CVD:

* chronic stable angina
* unstable angina
* uncomplicated myocardial infarction
* coronary artery bypass surgery
* percutaneous coronary angioplasty
* atherectomy or stent placement
* chronic stable angina pectoris
* stable Class I or Class II congestive heart failure
* stroke
* peripheral vascular disease

will be entered into the study if the CVD event or diagnosis occurred = 6 months ago.

Exclusion Criteria:

Patients with limited life expectancy (< 1 year) due to severe co-existing non-CVD disease such as:

* terminal illnesses such as terminal cancer
* CVD < 6 months ago
* Class III or IV CHF
* severe psychiatric illness such as psychosis
* manic depression
* alcohol abuse (> 21 drinks/week)
* serious chronic conditions like AIDS
* tuberculosis
* lupus
* and end-stage renal failure

will be excluded.

* Other exclusions include inability to understand English
* Lack of a landline telephone
* Unable to follow the study protocol
* Recent major surgery (< 3 months)
* Patients who are temporarily in the area and plan to move in < 1 year or will not be available for follow-up
* Those unable to provide informed consent.
* All patients excluded and reason for exclusion will be recorded.
* Prior to recruitment, each patient will be informed about the study and informed consent obtained.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 533 (Actual)
Dates: Start 2006-07; Primary Completion 2010-01 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Natarajan, MD MSc, Principal Investigator — VA New York Harbor Health Care System
Locations (1):
- VA New York Harbor Health Care System, New York, New York, United States

REFERENCES:
- [Result] Ulmer M, Robinaugh D, Friedberg JP, Lipsitz SR, Natarajan S. Usefulness of a run-in period to reduce drop-outs in a randomized controlled trial of a behavioral intervention. Contemp Clin Trials. 2008 Sep;29(5):705-10. doi: 10.1016/j.cct.2008.04.005. Epub 2008 May 6. PMID 18565801
- [Result] Friedberg JP, Lipsitz SR, Natarajan S. Challenges and recommendations for blinding in behavioral interventions illustrated using a case study of a behavioral intervention to lower blood pressure. Patient Educ Couns. 2010 Jan;78(1):5-11. doi: 10.1016/j.pec.2009.04.009. Epub 2009 Jun 13. PMID 19525084
- [Result] Friedberg JP, Rodriguez MA, Watsula ME, Lin I, Wylie-Rosett J, Allegrante JP, Lipsitz SR, Natarajan S. Effectiveness of a tailored behavioral intervention to improve hypertension control: primary outcomes of a randomized controlled trial. Hypertension. 2015 Feb;65(2):440-6. doi: 10.1161/HYPERTENSIONAHA.114.03483. Epub 2014 Nov 17. PMID 25403606
- [Derived] Rodriguez MA, Wang B, Hyoung S, Friedberg J, Wylie-Rosett J, Fang Y, Allegrante JP, Lipsitz SR, Natarajan S. Sustained Benefit of Alternate Behavioral Interventions to Improve Hypertension Control: A Randomized Clinical Trial. Hypertension. 2021 Jun;77(6):1867-1876. doi: 10.1161/HYPERTENSIONAHA.120.15192. Epub 2021 May 12. PMID 33979183

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage-matched Intervention (SM): 6 monthly phone calls of tailored counseling for diet, medication and exercise based on the Transtheoretical Model
- Health Education Intervention (HEI): 6 monthly phone calls of non-tailored counseling for diet, medication and exercise
- Usual Care (UC): treatment as usual with no additional counseling
Period: Overall Study
Arm/Group | Stage-matched Intervention (SM) | Health Education Intervention (HEI) | Usual Care (UC)
Started | 176 | 177 | 180
Completed | 156 | 159 | 170
Not Completed | 20 | 18 | 10
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Withdrawal by Subject | 6 | 2 | 0
Not completed — Lost to Follow-up | 12 | 14 | 6
Not completed — Moved out of state | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Stage-Matched Intervention (SMI): 6 monthly phone calls of tailored counseling for diet, medication and exercise based on the Transtheoretical Model
- Health Education Intervention (HEI): 6 monthly calls of nontailored counseling for diet, medication and exercise
- Usual Care (UC): treatment as usual for hypertension
- Total: Total of all reporting groups
Arm/Group | Stage-Matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC) | Total
Number analyzed (Participants) | 176 | 177 | 180 | 533
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age and Standard Deviation | 66.4 (8.8) | 66.5 (12.8) | 65.4 (10.2) | 66.1 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 7
  Male | 174 | 176 | 176 | 526
Race/Ethnicity, Customized [Number; unit: participants]
  White (non-Hispanic) | 81 | 60 | 71 | 212
  Black (non-Hispanic) | 65 | 77 | 70 | 212
  Hispanic | 24 | 29 | 29 | 82
  Other | 6 | 11 | 10 | 27
Marital status [Number; unit: participants]
  Married | 59 | 67 | 70 | 196
  Not Married | 117 | 110 | 110 | 337
Education [Number; unit: participants]
  High school graduate or below | 72 | 89 | 87 | 248
  Some college or higher | 104 | 88 | 93 | 285
Employment status [Number; unit: participants]
  Employed | 29 | 41 | 41 | 111
  Not employed | 147 | 136 | 139 | 422
Campus [Number; unit: participants]
  Manhattan campus | 96 | 96 | 97 | 289
  Brooklyn campus | 80 | 81 | 83 | 244
Smoking [Number; unit: participants]
  Current smoker | 35 | 32 | 32 | 99
  Current non-smoker | 141 | 145 | 148 | 434
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (5.2) | 31.2 (5.8) | 30.0 (4.8) | 30.5 (5.3)
Blood pressure control [Number; unit: participants] — Controlled BP was defined as systolic BP (SBP) less than130 mm Hg or Diastolic BP (DBP) less than 80 mm Hg in diabetes mellitus or chronic kidney disease, or SBP less than140 mm Hg or DBP less than 90 mm Hg in all others as per the BP guidelines at the time of the study.
  participants
    BP controlled | 75 | 72 | 80 | 227
    BP not controlled | 101 | 105 | 100 | 306
Diabetes Mellitus [Number; unit: participants] — From chart review
  participants
    Diabetes mellitus | 71 | 83 | 81 | 235
    No diabetes mellitus | 105 | 94 | 99 | 298
Ischemic Heart Disease (IHD) [Number; unit: participants] — self-reported
  participants
    History of IHD | 23 | 22 | 23 | 68
    No history of IHD | 153 | 155 | 157 | 465
History of revascularization [Number; unit: participants] — self-reported
  participants
    History of revascularization | 27 | 28 | 31 | 86
    No history of revascularization | 149 | 149 | 149 | 447
Hyperlipidemia [Number; unit: participants] — Hyperlipidemia was defined as LDL cholesterol of greater than or equal to 100 mg/dL from laboratory results
  participants
    Hyperlipidemia | 39 | 38 | 52 | 129
    No hyperlipidemia | 137 | 139 | 128 | 404
Estimated glomerular filtration rate (EGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 79.9 (25.5) | 83.2 (46.3) | 80.6 (28.4) | 81.3 (35.8)
Systolic Blood Pressure, mm Mg [Mean (Standard Deviation); unit: mm Hg] | 136.0 (11.8) | 137.2 (17.7) | 137.0 (12.9) | 136.7 (15.5)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 75.5 (9.3) | 76.1 (11.6) | 75.0 (11.1) | 75.5 (11.6)
Aerobic exercise [Mean (Standard Deviation); unit: hours per week] | 5.3 (8.1) | 4.5 (5.9) | 5.0 (6.7) | 4.9 (6.7)
Medication adherence by Morisky scale [Mean (Standard Deviation); unit: units on a scale] — Morisky medication-taking scale is a 4-item questionnaire scored from 0-4, with 4 being most adherent and less than 4 being considered nonadherent
  units on a scale | 3.4 (0.93) | 3.2 (0.67) | 3.3 (0.94) | 3.3 (0.88)
Number of antihypertensive medications [Mean (Standard Deviation); unit: medications] | 2.7 (1.5) | 2.8 (1.3) | 2.7 (1.3) | 2.7 (1.4)
Diet stage of change [Number; unit: participants] — The stages of change were: precontemplation, or no plans to adhere in <6 months; contemplation, or plans to adhere in 1-6 months; preparation, or plans to adhere within 1 month; action, or adherence for <6 months; and maintenance, or adherence for ≥ 6 months. Patients were considered adherent to diet if they reported eating the appropriate diet for hypertension (low in salt and fat with fruits, vegetables, and low-or non-fat dairy products) at least 6 days per week.
  participants
    Action or Maintenance | 69 | 67 | 70 | 206
    Precontemplation, Contemplation or Preparation | 107 | 110 | 110 | 327
Exercise Stage of Change [Number; unit: participants] — The stages of change were: precontemplation, or no plans to adhere in <6 months; contemplation, or plans to adhere in 1-6 months; preparation, or plans to adhere within 1 month; action, or adherence for <6 months; and maintenance, or adherence for ≥ 6 months. Exercise adherence was defined as self-reported aerobic exercise for at least 3 days per week for at least 20 minutes each time. We used the lower threshold for exercise adherence19, 20 due to our patient population with multiple comorbidities, consistent with Federal guidelines for older adults with chronic conditions.
  participants
    Action or Maintenance | 125 | 110 | 108 | 343
    Precontemplation, Contemplation, or Preparation | 51 | 67 | 72 | 190
Medication Stage of Change [Number; unit: participants] — The stages of change were: precontemplation, or no plans to adhere in <6 months; contemplation, or plans to adhere in 1-6 months; preparation, or plans to adhere within 1 month; action, or adherence for <6 months; and maintenance, or adherence for ≥ 6 months. Medication adherence was defined as self-report of taking BP medications as prescribed for at least 6 days per week.
  participants
    Action or Maintenance | 164 | 170 | 166 | 500
    Precontemplation, Contemplation or Preparation | 12 | 7 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Control
Description: Blood pressure Control at 6 months
Time Frame: 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
proportion of participants
  BP controlled | 0.646 | 0.543 | 0.458
  BP not controlled | 0.354 | 0.457 | 0.542
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI) vs Usual Care (UC); The study was an effectiveness trial of 2 active interventions, each compared with an active standard of care control group. We expected that 54% of patients on BP-lowering therapy would be properly controlled with HEI and 43% with UC, whereas we expected SMI to increase this to 69% control in 6 months. BP control and SBP were compared at 6 months across treatment arms using a 2.5% type I error (Bonferroni adjustment), ie, 1.25% for each of the 4 comparisons; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney) — BP control and SBP were compared at 6 months across treatment arms using a Bonferroni adjustment of 1.25% for each of the 4 comparisons (SMI versus UC and HEI versus UC for BP control and SBP separately). This p-value is for comparison of SMI vs. UC
Statistical Analysis 2: Comparison: Health Education Intervention (HEI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.108, Wilcoxon (Mann-Whitney) — BP control and SBP were compared at 6 months across treatment arms using a Bonferroni adjustment of 1.25% for each of the 4 comparisons (SMI versus UC and HEI versus UC for BP control and SBP separately). This p-value is for comparison of HEI vs. UC

2. Primary Outcome: Systolic Blood Pressure
Description: Mean systolic Blood Pressure
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
mm Hg | 131.2 [129.1 to 133.3] | 131.8 [129.9 to 133.7] | 134.7 [132.7 to 136.7]
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI) vs Usual Care (UC); The study was designed as an effectiveness trial of 2 active interventions, each compared with an active standard of care control group. The study was not powered to test comparisons between the 2 active intervention arms; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney) — BP control and SBP were compared at 6 months across treatment arms using a 2.5% type I error (Bonferroni adjustment), 1.25% for each of the 4 comparisons (SMI versus UC and HEI vs UC for BP control and SBP separately). This p-value is for SMI vs UC
Statistical Analysis 2: Comparison: Health Education Intervention (HEI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney) — BP control and SBP were compared at 6 months across treatment arms using a Bonferroni adjustment of 1.25% for each of the 4 comparisons (SMI versus UC and HEI vs UC for BP control and SBP separately). This p-value is for comparison of HEI vs. UC

3. Secondary Outcome: Change in Proportion With BP Under Control From Baseline to 6 Months
Time Frame: 6 months
Measure: Number; unit: Proportion of participants
Groups:
- Health Education Intervention (HEI): 6 monthly phone calls of nontailored counseling for diet, medication and exercise
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
Proportion of participants | .197 | .118 | .019
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI); Test type: Superiority or Other; p < 0.000003, McNemar — Change in BP control were compared by treatment arm using a 1.67% type I error (with Bonferroni adjustment), ie, 1.67% for each assessment of change in proportion with BP under control from baseline to 6 months by SMI, HEI or UC (3 tests)
Statistical Analysis 2: Comparison: Health Education Intervention (HEI); Test type: Superiority or Other; p = 0.012, McNemar — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Usual Care (UC); Test type: Superiority or Other; p = 0.89, McNemar — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to 6 Months
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Stage-matched Intervention (SMI): 6 monthly calls targeting diet, medication and exercise adherence tailored using the Transtheoretical Model
- Health Education Intervention (HEI): 6 monthly calls of non-tailored education about diet, medication and exercise recommendations
- Usual Care (UC): Treatment as usual for hypertension with no counseling
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
mm Hg | -4.7 [-6.9 to -2.5] | -5.4 [-8.5 to -2.3] | -2.7 [-5 to -0.4]
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI); Test type: Superiority or Other; p < 0.009, Wilcoxon (Mann-Whitney) — Change in SBP were compared by treatment arm using a 1.67% type I error (Bonferroni adjustment), ie, 1.67% for each of the 3 comparisons by arm (6-month-baseline for SMI, HEI and UC separately)
Statistical Analysis 2: Comparison: Health Education Intervention (HEI); Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Usual Care (UC); Test type: Superiority or Other; p = 0.9, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 4, analysis 1]

5. Secondary Outcome: Change in Number of Cardio Exercise Hours From Baseline to 6 Months
Time Frame: baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
hours | -0.29 [-1.7 to 1.1] | 0.53 [-0.6 to 1.7] | -0.43 [-1.4 to 0.6]
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.880, Wilcoxon (Mann-Whitney) — Since we are performing 3 tests, we will adjust the type I error to 0.017
Statistical Analysis 2: Comparison: Health Education Intervention (HEI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.318, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: Change in Morisky Score From Baseline to 6 Months
Description: Morkisy medication adherence self-report questionnaire, a 4-item questionnaire scored from 0-4. A score of 4 is considered most adherent, and scores of less than 4 are defined as nonadherent
Time Frame: baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Health Education Intervention (HEI): 6 months of non-tailored counseling for diet, medication and exercise
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
units on a scale | 0.25 [0.1 to 0.4] | 0.25 [0.1 to 0.4] | 0.14 [0 to 0.3]
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.306, Wilcoxon (Mann-Whitney) — Since we are performing 3 tests, we will adjust the type I error to 0.017
Statistical Analysis 2: Comparison: Health Education Intervention (HEI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.205, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Diet Stage of Change
Description: The stages of change were: precontemplation, or no plans to adhere in <6 months; contemplation, or plans to adhere in 1-6 months; preparation, or plans to adhere within 1 month; action, or adherence for <6 months; and maintenance, or adherence for ≥ 6 months. Patients were considered adherent to diet if they reported eating the appropriate diet for hypertension (low in salt and fat with fruits, vegetables, and low-or non-fat dairy products) at least 6 days per week.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Usual Care (UC): treatment as usual
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
participants
  Action or Maintenance | 87 | 73 | 73
  Precontemplation, Contemplation or Preparation | 69 | 86 | 97
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.011, Chi-squared — Since we are performing 3 tests, we will adjust the type I error to 0.017
Statistical Analysis 2: Comparison: Health Education Intervention (HEI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.638, Chi-squared — Since we are performing 3 tests, we will adjust the type I error to 0.017

8. Secondary Outcome: Exercise Stage of Change
Description: The stages of change were: precontemplation, or no plans to adhere in <6 months; contemplation, or plans to adhere in 1-6 months; preparation, or plans to adhere within 1 month; action, or adherence for <6 months; and maintenance, or adherence for ≥ 6 months. Exercise adherence was defined as self-reported aerobic exercise for at least 3 days per week for at least 20 minutes each time. We used the lower threshold for exercise adherence due to our patient population with multiple comorbidities, consistent with Federal guidelines for older adults with chronic conditions.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
participants
  Action or Maintenance | 128 | 124 | 126
  Precontemplation, Contemplation or Preparation | 28 | 35 | 44
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.012, Chi-squared — Since we are performing 3 tests, we will adjust the type I error to 0.017
Statistical Analysis 2: Comparison: Health Education Intervention (HEI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.333, Chi-squared — Since we are performing 3 tests, we will adjust the type I error to 0.017

9. Secondary Outcome: Medication Stage of Change
Description: The stages of change were: precontemplation, or no plans to adhere in <6 months; contemplation, or plans to adhere in 1-6 months; preparation, or plans to adhere within 1 month; action, or adherence for <6 months; and maintenance, or adherence for ≥ 6 months. Medication adherence was defined as self-report of taking BP medications as prescribed for at least 6 days per week.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Number analyzed (Participants) | 156 | 159 | 170
participants
  Action or Maintenance | 148 | 156 | 163
  Precontemplation, Contemplation or Preparation | 8 | 3 | 7
Statistical Analysis 1: Comparison: Stage-matched Intervention (SMI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.581, Chi-squared — Since we are performing 3 tests, we will adjust the type I error to 0.017
Statistical Analysis 2: Comparison: Health Education Intervention (HEI) vs Usual Care (UC); Test type: Superiority or Other; p = 0.502, Chi-squared — Since we are performing 3 tests, we will adjust the type I error to 0.017

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Stage-matched Intervention (SMI) | Health Education Intervention (HEI) | Usual Care (UC)
Serious Adverse Events (participants affected / at risk) | 3/176 | 1/177 | 3/180
Other Adverse Events (participants affected / at risk) | 14/176 | 7/177 | 9/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage-matched Intervention (SMI) (N=176) | Health Education Intervention (HEI) (N=177) | Usual Care (UC) (N=180)
Heart attack (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage-matched Intervention (SMI) (N=176) | Health Education Intervention (HEI) (N=177) | Usual Care (UC) (N=180)
Angina (Cardiac disorders) | 5 (5) | 3 (3) | 4 (4)
broken bones (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 1 (1)
torn ligament (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
hypertensive emergency (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Coronary artery bypass graft (Surgical and medical procedures) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes